CLINICAL TRIAL: NCT01865058
Title: The Use of 18 F-FDG Positron Emission Tomography (PET) in the Early Response Evaluation of Diffuse Large B-cell Lymphoma.
Brief Title: The Use of PET for the Early Response Evaluation in Patients With Diffuse Large B-cell Lymphoma.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Karen Juul Mylam, MD, Odense University Hospital
Other Study IDs: DLG-PET 10.06
Record Dates: First submitted 2013-05-01; First posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DLBCL: Patients with newly diagnosis of diffuse large B-cell lymphoma is offered enrollment in this protocol.

SUMMARY:
Non-Hodgkin lymphoma (NHL) is one of the more frequent cancers in the western world with approx. 800 new cases annually in Denmark. Diffuse large B-cell lymphoma (DLBCL) in Denmark accounts for almost 40% of newly diagnosed NHL cases. Treatment with the combination of chemotherapy and monoclonal antibodies has significantly improved prognosis over the past decade, but a large proportion of patients with DLBCL will continue to relapse with our current treatment options. Therefore, there is a need for reliable methods for detection of treatment response as early as possible in the treatment course in order to identify patients who respond poorly to standard treatment and potentially would benefit from a change in treatment strategy. This has still not been established, but a valid early marker is required in order to allow randomized trials of treatment stratified by early response. One of the most promising applications of PET is the metabolic assessment of the early response of cancer treatment.

This study is a national prospective multicenter study emanating from the Danish Lymphoma Group (DLG). Patients are scanned after each of the early 4 cycles of chemo therapy. The aim is to establish the correct timing of response evaluation. Additionally, the investigators wish to investigate the optimal qualitative and quantitative method of response assessment in order to predict post-therapeutic remission and long-term prognosis.This study will contribute to interim-PET being implemented in the most optimal way in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

-Age>18 years

Exclusion Criteria:

* Previously treatment with chemotherapy or irradiation
* Primary CNS lymphoma
* Recurrent lymphoma
* Transformation from indolent lymphoma
* Presence of diabetes mellitus, HIV, chronic inflammatory disease or infections
* Planned for curative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosis of Diffuse Large B-cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-02 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
Progression free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 2 years, 3 years

OTHER OUTCOMES:
Treatment response (CR, PR, PD) | Up to 24 weeks
  The time frame is from baseline PET scanning to completions of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Juul Mylam, MD, Principal Investigator — Hematology research Unit, Odense University Hospital
Locations (1):
- Hematology Rearch Unit, Odense University Hospital, Odense, Fyn, Denmark